CLINICAL TRIAL: NCT00599677
Title: Randomized Controlled Trial of Acupuncture for Functional Dyspepsia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2006CB5045012; 2006CB5045012
Record Dates: First submitted 2008-01-04; First posted 2008-01-24 (Estimated); Last update posted 2011-11-09 (Estimated); Status verified 2011-11

CONDITIONS: Functional Dyspepsia
Keywords: acupuncture; meridian; acupoint
MeSH Terms: interventions — Acupuncture Therapy; itopride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- group 1 (Experimental): specific acupoints of Stomach meridians
  Interventions: Other: acupuncture
- group 2 (Experimental): Non-specific acupoints of Stomach meridians
  Interventions: Other: acupuncture
- group 3 (Experimental): alarm and transport points
  Interventions: Other: acupuncture
- group 4 (Experimental): acupoints of the other meridian
  Interventions: Other: acupuncture
- group 5 (Sham Comparator): non-acupoints
  Interventions: Other: acupuncture
- group 6 (Active Comparator): Itopride
  Interventions: Drug: Itopride

INTERVENTIONS:
Other: acupuncture — Subjects are treated five days a week continuously, and for four weeks.They are treated 30min every time.
  Arms: group 1; group 2; group 3; group 4; group 5
Drug: Itopride — Each pill weighs 50mg, once a pill, three times a day. The pills are taken half an hour before meals, and be taken 4 weeks continuously.
  Other Names: Itopride Hydrochloride Tablets
  Arms: group 6

SUMMARY:
The purpose of the study is to testify the efficacy of treating functional dyspepsia with acupuncture, and provide evidence for the hypothesis that "Acupuncture effect is based on meridians, and gathering of meridian Qi is the key point."

DETAILED DESCRIPTION:
The purpose of the study is to testify whether acupuncture is effective for functional dyspepsia, through treating functional dyspepsia patient for a month, using different acupoints according to literatures of treating migraine with acupuncture, and using Itopride as controlled group, and try to provide clinical evidence for the hypothesis that"Acupuncture effect is based on meridians, and gathering of meridian Qi is the key point."

ELIGIBILITY:
Inclusion Criteria:

1. Consistent with the diagnostic criteria of functional dyspepsia.
2. Age of a subject is older than 18 and is younger than 65.（including 18 and 65）
3. Did not take any gastroenteric dynamic drugs in the last 15 days, and did not take part in any clinical trial.
4. Informed consent is signed by a subject or his lineal relation.

Exclusion Criteria:

1. Patients with any contraindications of Itopride.
2. Patients who are unconscious, psychotic.
3. Patients with aggravating tumor and other serious consumptive disease, and who are subject to infection and bleeding.
4. With serious protopathy or disease of cardiovascular, liver, renal, gastrointestinal, hematological systems and so on.
5. Pregnant women or women in lactation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 720 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Nepean Dyspepsia Index | 4 weeks

SECONDARY OUTCOMES:
Symptoms Index of Dyspepsia | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fan-rong Liang, master, Study Chair — Chengdu University of TCM
Locations (1):
- Chengdu University of TCM, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Ma T, Zeng F, Li Y, Wang CM, Tian X, Yu S, Zhao L, Wu X, Yang M, Wang D, Liang F. Which subtype of functional dyspepsia patients responses better to acupuncture? A retrospective analysis of a randomized controlled trial. Forsch Komplementmed. 2015;22(2):94-100. doi: 10.1159/000380983. Epub 2015 Mar 11. PMID 26021959
- [Derived] Zhao L, Zhang FW, Li Y, Wu X, Zheng H, Cheng LH, Liang FR. Adverse events associated with acupuncture: three multicentre randomized controlled trials of 1968 cases in China. Trials. 2011 Mar 24;12:87. doi: 10.1186/1745-6215-12-87. PMID 21435214
- [Derived] Zheng H, Tian XP, Li Y, Liang FR, Yu SG, Liu XG, Tang Y, Yang XG, Yan J, Sun GJ, Chang XR, Zhang HX, Ma TT, Yu SY. Acupuncture as a treatment for functional dyspepsia: design and methods of a randomized controlled trial. Trials. 2009 Aug 23;10:75. doi: 10.1186/1745-6215-10-75. PMID 19698147